CLINICAL TRIAL: NCT02866968
Title: Clinical Outcomes of Femtosecond Laser-assisted Pterygium Surgery (FLAPS)
Acronym: FLAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Eye Research Institute (Other)
Responsible Party: Principal Investigator, Jodhbir Mehta, Prof, Singapore Eye Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R1361/47/2016
Record Dates: First submitted 2016-07-19; First posted 2016-08-15 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Femtosecond Laser-assisted Pterygium Surgery (FLAPS) (Experimental): All patients included will undergo FLAPS in one eye.
  Interventions: Procedure: FLAPS

INTERVENTIONS:
Procedure: FLAPS — Surgical procedures will involve 1) excision of pterygium tissue from cornea and conjunctiva, 2) resection of residual Tenon and coagulation to stop any bleeding 3) preparation of a 8x8 mm conjunctiva autograft in the superior bulbar conjunctiva with the femtosecond laser (12 o´clock position) and 4) fixation of the graft with fibrin glue to the resection site.

SUMMARY:
The study will be a pilot interventional case series aiming to treat 30 patients with Femtosecond Laser-assisted Pterygium Surgery (FLAPS). All patients included will undergo FLAPS in one eye. All procedures will be performed in SNEC by fully qualified surgeons. The doctor is informed of the procedure on the day of.

ELIGIBILITY:
Inclusion Criteria:

* A pterygium will be defined as a wing-shaped growth of fibrotic connective tissue onto the cornea originating from the nasal conjunctiva.
* Only patients older than 21 years will be included.
* No gender criteria are applied.
* Only individuals with the mental capacity to provide informed consent will be included.

More specifically, all the following inclusion criteria must be met:

* Patients have primary pterygium encroaching onto the cornea by a minimum of 1 mm.
* Patients are willing and able to sign a written Informed Consent Form prior to any study-specific procedures.
* Patients are willing and able to return for scheduled follow-up examinations for 12 months after the surgery.

Exclusion Criteria:

* Patients with prior history of pterygium surgery.
* Patients with a prior history of glaucoma filtration surgery.
* Patients with optic atrophy.
* Patients with ocular pathology or disease that might confound the outcome or increase the risk of adverse events.
* Patients with a prior history of vitrectomy.
* Patients with central corneal scarring.
* Patients with residual, recurrent, active or uncontrolled eyelid disease.
* Patients with any conjunctival scarring other than pterygium, that could affect surgery outcome.
* Patients with anterior segment pathology.
* Patients with any corneal abnormality.
* Patients with any progressive retinal disease or subjects with a history or evidence of retinal vascular occlusion and/or hypercoagulability, because of the risks associated with high pressures during suction application.
* Patients with amblyopia or strabismus or those who are at risk for developing strabismus postoperatively as determined by corneal light reflex and cover-uncover testing.
* Patients who are pregnant, lactating, of child-bearing potential and not practising a medically approved method of birth control, or planning to become pregnant during the course of the trial, and patients with other conditions associated with fluctuation of hormones that could lead to refractive changes.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of FLAPS | 12 month follow-up
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Recurrence free survival over 12 months. | 12 month follow-up
  Number of cases with pterygium recurrence during 12 month follow-up
Visual acuity | Day 0, 7 and 1, 3, 6, 12 months
  Best-spectacle corrected visual acuity (BSCVA) to be measured with a Snellen chart at 6 meters, then converted to logarithmic minimum angle of resolution unit to allow for averaging and statistical analysis
Refraction | Day 0, 7 and 1, 3, 6, 12 months
  Non-invasive non-contact measurement with autorefractor measured in spherical and cylindrical diopters
Corneal Topography | (Day 0, 7 and 1, 3, 6, 12 months)
  Non-invasive non-contact scan with OCULUS Pentacam, measurement of cylindrical diopters

CONTACTS AND LOCATIONS:
Overall Officials: Jodhbir S Mehta, Prof, Principal Investigator — Singapore Eye Research Institute
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

REFERENCES:
- [Derived] Ting DSJ, Liu YC, Lee YF, Ji AJS, Tan TE, Htoon HM, Mehta JS. Cosmetic outcome of femtosecond laser-assisted pterygium surgery. Eye Vis (Lond). 2021 Mar 6;8(1):7. doi: 10.1186/s40662-021-00230-w. PMID 33673873